CLINICAL TRIAL: NCT03626805
Title: Muscle Tenderness and Hardness in Migraine Patients
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Jeppe Hvedstrup Mann, PhD Student, Danish Headache Center
Other Study IDs: 001
Record Dates: First submitted 2018-06-05; First posted 2018-08-13 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Migraine Disorders; Muscle Tenderness; Headache Disorders, Primary; Nervous System Diseases; Headache, Migraine
MeSH Terms: conditions — Migraine Disorders; Myalgia; Headache Disorders, Primary; Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraine patients: Migraine patients attending the Danish Headache Centre
- Healthy Controls: Age and sex matched

SUMMARY:
The aim of the study is to examine symptomatology, quantitative sensory test (QST) parameters, muscle tenderness and muscle hardness in migraine patients interictally and compare with healthy controls

DETAILED DESCRIPTION:
Migraine patients exhibit different symptomatology and responses to treatment. For example do many migraine patients have neck symptoms, despite they apparently do not have any neck disorders.Furthermore the response to treatment differs between patients. Differences in symptomatology, QST parameters and muscle stiffness can be used to subdivide and phenotype migraine patients.

The investigators are examining migraine patients with:

A semistructured interview, Quantitative sensory testing (cold pain threshold, heat pain threshold and Pin Prick), Muscle tenderness (total tenderness score, local tenderness score and stimulus response curve), and muscle hardness with ultrasound elastography. All tests are performed the same day

ELIGIBILITY:
Inclusion Criteria:

* Migraine Patients from the Danish Headache Centre. Migraine classified using the International Classification of Headache Disorders (ICHD3) criteria.

Exclusion Criteria:

* Pregnant or lactating women
* Musculoskeletal injuries in the neck or shoulder
* Other primary headache disorders than migraine or Tension Type Headache
* On the time of examination: Migraine free for at least 48 hours
* On the time of examination: haven't trained the upper body for at least 48 hours
* On the time of examination: haven't used painkillers for at least 48 hours

Healthy controls:

Exclusion Criteria:

* Pregnant or lactating women
* Musculoskeletal injuries in the neck or shoulder
* Migraine disorders
* 1. degree relatives with migraine disorders
* Over 1 day of tension type headache a month.
* On the time of examination: haven't trained the upper body for at least 48 hours
* On the time of examination: haven't used painkillers for at least 48 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migraine patients are recruited from the out-patient clinic at the Danish Headache Center.
  Healthy controls are recruited through web-sites.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-08-13 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Logistic regression model, Neck Stiffness | 3 hours
  We would like to examine the relationship between the variable variable: Neck stiffness during migraine attack (Yes/No) and the Independent variables: Total Tenderness Score (summed score from 8 points bilateral, each point can score 0-3), Migraine localisation (occipital: Yes/No), Tension Type Headache, Allodynia (yes/No), Stimulus response curve (Pressure and Pain).
  The result shows how much of the variability in neck stiffness that can be explained by the independent variables.
Pericranial Muscle Tenderness | 3 hours
  We will examine whether patients with neck stiffness during migraine attack (yes/no) have higher tenderness scores compared to patients without neck stiffness during migraine attacks, when correcting for headache frequency.
Muscle Hardness measured by ultrasound elastography | 3 hours
  Muscle hardness (m/s) in migraine patients compared to healthy controls.corrected for age, BMI and sex
Muscle hardness measured by ultrasound elastography in migaine patients | 3 hours
  Muscle hardness (m/s) in migraine patients with neck stiffness during migraine attacks compared to migraine patients without neck stiffness during migraine attacks. Corrected for age, BMI and sex.

SECONDARY OUTCOMES:
Multiple Regression model, Total Tenderness Score | 3 hours
  We would like to examine the relationship between the dependent variable: Total Tenderness Score(summed score from 8 points bilateral, each point can score 0-3), and the Independent variables: Neck Pain in general(Yes/No), Migraine localisation (occipital: Yes/No), Headache Frequency(days/month), Allodynia (Yes/No), Years with Migraine(Number of years)
Logistic regression model, Neck pain in general | 3 hours
  We would like to examine the relationship between the variable variable: Neck pain in general (Yes/No) and the independent variables: Tension Type Headache(yes/no), Migraine localisation, Headache Frequency(Headache days/month), Allodynia(yes/No), Years with Migraine(number of years)
Next migraine attack, Cox proportional hazards model | 3 hours
  Using the prospective diary, we will examine the relationship between pericranial muscle tenderness and the next migraine attack, when correcting for headache frequency

OTHER OUTCOMES:
Correlation analysis of muscle hardness and headache frequency | 3 hours
  Muscle hardness will be measured with ultrasound elastography. Headache frequency is self-reported
Correlation analysis of muscle hardness and muscle tenderness assessed with the total tenderness score. | 3 hours
  Muscle hardness will be measured with ultrasound elastography.
Correlation analysis of muscle hardness and pressure pain threshold assessed with an pressure algometer. | 3 hours
  Muscle hardness will be measured with ultrasound elastography

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe H Mann, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hvedstrup J, Kolding LT, Ashina M, Schytz HW. Increased neck muscle stiffness in migraine patients with ictal neck pain: A shear wave elastography study. Cephalalgia. 2020 May;40(6):565-574. doi: 10.1177/0333102420919998. Epub 2020 Apr 15. PMID 32295400